CLINICAL TRIAL: NCT05676138
Title: Pharmacokinetics and Pharmacodynamics of Multidrug-regimens for Mycobacterium Abscessus Pulmonary Disease
Brief Title: PK and PD of Antibiotics for Treatment of Mycobacterium Abscessus Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Joon Yim, Professor, Seoul National University Hospital
Other Study IDs: 2017-2154
Record Dates: First submitted 2022-12-08; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Nontuberculous Mycobacterial Pulmonary Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measuring PK and PD indices in patients who receive conventional treatment — Measuring plasma concentration of commonly used antibiotics in NTM-PD

SUMMARY:
Investigating the PK and PD indices in patients with M. abscessus complex-PD who will be treated with a currently recommended regimen, minimum inhibitory concentrations of organism, and their relation with clinical outcomes

DETAILED DESCRIPTION:
Nontuberculous mycobacteria (NTM), consisting of more than 200 mycobacteria other than M. tuberculosis and M. leprae, is an environmental organism, which can be isolated from soil, dust and water. NTM can cause chronic diseases in human and the most common manifestation is pulmonary disease (PD) . During the last decades, the burden of NTM-PD in rapidly increasing in global. In South Korea, the incidence has increased from 1.0 per 100,000 population in 2003 to 17.9 per 100,00 population in 2016.

M. abscessus complex is a group of rapidly growing mycobacteria (RGM). M. abscessus complex can be divided into three subspecies: M. abscessus subspecies abscessus (hereafter, referred to as M. abscessus), M. abscessus subspecies massiliense (M. massiliense), and M. abscessus subspecies bolletii (M. bolletii). Among the RGMs, M. abscessus complex is the most common pathogen for respiratory infection. With its distinctive surface properties and type VII secretion system (ESX-4), M. abscessus complex can cause progressive infection in patients with structural lung diseases such as cystic fibrosis.

Treatment of M. abscessus complex is extremely difficult. M. abscessus complex is generally resistant to most classes of antibiotics due to decreased cell wall permeability, induction of efflux pumps, and modification of drug targets. Especially, the presence of function erm(41) gene in M. abscessus confers inducible resistance to macrolide, which is the core drug of NTM-PD. As a result, multidrug regimens including at least three or four active drugs based on in vitro susceptibility are recommended for M. abscessus complex-PD.

Even though these complex and intensified treatments are administered in real clinical practice, the optimal drugs, dosage and duration of therapy are still not understood. Moreover, treatment outcomes are still unsatisfactory. According to the dataset from 303 patients with M. abscessus complex-PD, the treatment success rates were 33.0% for M. abscessus and 56.7% for M. massiliense, respectively. The unfavorable outcomes of currently recommended regimens are partly explained by an incomplete understanding of the relationship between pharmacokinetics (PK) of drugs used, in vitro susceptibility and treatment outcomes. To improve treatment outcomes, it should be preceded to figure out the potential efficacy of currently recommended regimens for M. abscessus complex-PD.

This will be performed as a prospective pharmacokinetic study for patients with M. abscessus complex-PD. Patients, who are scheduled to initiate treatment for M. abscessus complex-PD between 1 January 2023 and 31 December 2024 at Seoul National University Hospital, will be the subject of study. The size of population is estimated to be 40.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years old or more
* Fulfilling the criteria of NTM-PD (1, 13), for which causative organism belongs to M. abscessus or M. massiliense
* Needing a new antibiotic treatment for M. abscessus complex-PD due to symptomatic aggravation, radiographic progression or both (those who have previous history of treatment are eligible)
* Consenting to receive antibiotic treatment based on currently recommended regimens (1, 13) and to participate in this study

Exclusion Criteria:

* Receiving any treatment for NTM-PD within 4 weeks
* Having end-stage renal disease needing hemodialysis, chronic liver disease, or active malignancy needing treatment during the treatment period

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with M. abscessus pulmonary disease, who receive conventional antibiotic treatment based on the currently recommended guideline.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | 2 weeks of treatment
  Cmax of guideline-recommended antibiotics in patients will be measured
Time to Cmax | 2 weeks of treatment
  Time to Cmax of guideline-recommended antibiotics in patients will be measured
Area under the curve from 0 to 24 hours after dosing | 2 weeks of treatment
  AUC24 of guideline-recommended antibiotics in patients will be measured
Plasma half-life | 2 weeks of treatment
  Plasma half-life of guideline-recommended antibiotics in patients will be measured

SECONDARY OUTCOMES:
Time to culture positivity (days) by AUC24 (mg x h/L) | 2 weeks of treatment
  Time to culture positivity (mycobacterial culture in liquid media) from sputum represents the effect of treatment. The time to culture positivity (days) from sputum collected at 2 weeks of treatment will be measrued according to AUC24.
Time to culture positivity (days) by Cmax (mg /L) | 2 weeks of treatment
  Time to culture positivity (mycobacterial culture in liquid media) from sputum represents the effect of treatment. The time to culture positivity (days) from sputum collected at 2 weeks of treatment will be measrued according to Cmax.

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: Undecided